CLINICAL TRIAL: NCT06463288
Title: Comparison of Jacobson Relaxation Technique and Pranayama Technique in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/ 31831 Iqra
Record Dates: First submitted 2024-03-04; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: COPD; Shortness of Breath; Quality of Life; Cough
Keywords: COPD; Jacobson Technique; Pranayama Technique; SOB
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Cough

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jacobson's Technique (Experimental): Participant in the group A were instructed to perform the Jacobson relaxation technique.
  * Quite place were chosen where there is no disturbance.
  * Patients were relax either on the lying position or sitting position with head well-supported.
  * Patients were instructed to loosen any tight clothing.
  * Patients were educated for muscles of each group emphasis on attention on that muscle group only.
  * Repeat this three times, constrict the muscle and then relax, tens the muscle and maintain it for five seconds then relax it lightly and then tense and relax. Constrict the muscle very slightly then relax it. Focus on each muscle group and then decide to relax the target muscle.
  Interventions: Procedure: Jacobsons Breathing Technique
- Pranayama Technique (Active Comparator): Participant in group B were instructed to perform the pranayama relaxation technique.
  * Quite place were chosen where there is no disturbance and patient were relaxed in sitting position with spine straight.
  * In this technique patients were instructed to perform different type of pranayama techniques.
  * Guide the participants to take a steady breath in through your both nostrils. Then inhale until you reach your total lung capacity, maintaining a tall spine.
  Treatment was continuous 4 weeks, 3 times in a week for 15 mint. Assessment was done through the tool before and after the treatment.
  Interventions: Procedure: Pranayama Technique

INTERVENTIONS:
Procedure: Jacobsons Breathing Technique — Quality of life, cough and sputum analysis, spirometry, and shortness of breath were assessed.
  Arms: Jacobson's Technique
Procedure: Pranayama Technique — Quality of life, cough and sputum analysis, spirometry, and shortness of breath were assessed.
  Arms: Pranayama Technique

SUMMARY:
Comparison of Jacobson Relaxation Technique and Pranayama Technique in patients with COPD

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease is a chronic inflammatory lung disease that cause obstructed airflow from the lungs. Symptoms include Breathing difficulty. cough, mucus production and wheezing. Its typically caused by long term exposure to irritating gasses or particulate matter, most often from cigarette smoker. in this study we compare the effect of Jacobson relaxation technique and Pranayama technique on the SOB, Cough, sputum and quality of life in COPD patients.

Data were collected from Gulab Devi Chest Hospital, General Hospital, Jinnah Hospital and Mayo Hospital Lahore. Data were collected by the lottery method. Borg dyspnea scale, Spirometry, CASA-Q and Quality of life questionnaire were used before and after the intervention. Treatment was continuous 4 weeks, 3 times in a week for 15 mint. Assessment was done through the tool before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* • Patients of Age between 40 and 70.

  * Both Genders (Male, Female) were included.
  * Stage 2 patient with COPD with Dyspnea FEV1 <70% and Maximal Expiratory Pressure = 50% (Gold Criteria) were included.
  * Cognitive Stable patients were included.
  * Those Patients were included who were clinically stable without exacerbations in the past 01 month.

Exclusion Criteria:

* • Common Cough

  * Upper respiratory tract inflammation
  * Patients who have other co-morbid diseases which prevents them from exercise training, for example, disability due to neurological, orthopedic and acute cardiac causes
  * Patients who were mentally and physically and sick to join at the hospital or research site for training
  * Patients who were already participated or completed or in a P.R program in the past one year.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Dyspnea Severity (Borg Scale) | 4 weeks
  The Borg scale measures the severity of dyspnea (shortness of breath).
  Scale Details:
  Full Title: Borg Rating of Perceived Exertion (RPE) ScaleFull Title: Borg Rating of Perceived Exertion (RPE) Scale Minimum Value: 0 (No breathlessness at all) Maximum Value: 10 (Maximal breathlessness) Interpretation: Higher scores indicate worse outcomes, meaning greater severity of dyspnea.
Cough and Sputum Analysis (CASA-Q) | 4 Weeks
  The CASA-Q (Cough and Sputum Assessment Questionnaire) evaluates the severity and impact of cough and sputum production.
  Scale Details:
  Full Title: Cough and Sputum Assessment Questionnaire (CASA-Q) Minimum Value: 0 (No symptoms) Maximum Value: 100 (Severe symptoms) Interpretation: Higher scores indicate worse outcomes, meaning more severe symptoms of cough and sputum.
Spirometry (FEV1 and FVC) | 4 Weeks
  Spirometry will be used to measure lung function, specifically Forced Expiratory Volume in 1 second (FEV1) and Forced Vital Capacity (FVC).
  Scale Details:
  Full Title: Spirometry (FEV1 and FVC) Minimum Value: Variable (dependent on patient's lung function) Maximum Value: Variable (dependent on patient's lung function) Interpretation: Higher values typically indicate better lung function.

SECONDARY OUTCOMES:
Quality of Life (SF-36 Questionnaire) | 4 Weeks
  The SF-36 (Short Form Health Survey) questionnaire assesses the overall quality of life.
  Scale Details:
  Full Title: SF-36 Health Survey Minimum Value: 0 (Worst possible health state) Maximum Value: 100 (Best possible health state) Interpretation: Higher scores indicate better quality of life.
Patient Satisfaction (Patient Satisfaction Questionnaire) | 4 Weeks
  The Patient Satisfaction Questionnaire measures the satisfaction of patients with the treatment they received.
  Full Title: Patient Satisfaction Questionnaire (PSQ) Minimum Value: 1 (Very dissatisfied) Maximum Value: 5 (Very satisfied) Interpretation: Higher scores indicate greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Sumera Hameed, MS, Principal Investigator — Riphah International University
Locations (1):
- Gulab Devi Chest Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pauwels RA, Buist AS, Ma P, Jenkins CR, Hurd SS; GOLD Scientific Committee. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: National Heart, Lung, and Blood Institute and World Health Organization Global Initiative for Chronic Obstructive Lung Disease (GOLD): executive summary. Respir Care. 2001 Aug;46(8):798-825. No abstract available. PMID 11463370
- [Background] Petty TL. The history of COPD. Int J Chron Obstruct Pulmon Dis. 2006;1(1):3-14. doi: 10.2147/copd.2006.1.1.3. PMID 18046898
- [Background] Ozgundondu B, Gok Metin Z. Effects of progressive muscle relaxation combined with music on stress, fatigue, and coping styles among intensive care nurses. Intensive Crit Care Nurs. 2019 Oct;54:54-63. doi: 10.1016/j.iccn.2019.07.007. Epub 2019 Jul 29. PMID 31371164
- [Background] Ranjita R, Hankey A, Nagendra HR, Mohanty S. Yoga-based pulmonary rehabilitation for the management of dyspnea in coal miners with chronic obstructive pulmonary disease: A randomized controlled trial. J Ayurveda Integr Med. 2016 Jul-Sep;7(3):158-166. doi: 10.1016/j.jaim.2015.12.001. Epub 2016 Aug 18. PMID 27545747
- [Background] Basoglu OK, Atasever A, Bacakoglu F. The efficacy of incentive spirometry in patients with COPD. Respirology. 2005 Jun;10(3):349-53. doi: 10.1111/j.1440-1843.2005.00716.x. PMID 15955148